CLINICAL TRIAL: NCT07034820
Title: Double-Blind, Placebo-Controlled, Parallel-Group Randomized Controlled Trial to Evaluate the Efficacy and Safety of Nimsai Herbal in Patients With Grade 2-3 Hemorrhoids
Brief Title: War-Drill Model Guided Treatment of Hemorrhoids With Nimsai Herbal (NAJ)
Acronym: NAJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nimsai Academia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA-2024-01
Record Dates: First submitted 2025-06-16; First posted 2025-06-24 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Hemorrhoids; Hemorrhoidal Disease
Keywords: Hemorrhoids; Hemorrhoidal Disease; Pathogenesis; War-Drill Model; Sine Qua Non Hypothesis; Venous Congestion; Nimsai Herbal; Randomized Controlled Trial; Clinical Trial; Treatment; Early Diagnosis; Biological Early-Warning System; Inflammatory Bowel Disease; Anal Fissure; Rectal Polyps; Hormonal Fluctuations; Parola Phenomenon; Systemic Therapy; Gastroenterology
MeSH Terms: conditions — Hemorrhoids; Hyperemia; Disease; Inflammatory Bowel Diseases; Fissure in Ano

STUDY DESIGN:
Intervention Model Description: Participants were randomized to either the Nimsai Herbal group or the placebo group, with both groups receiving treatment concurrently.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study employed a robust double-blind design where the Nimsai Herbal and placebo treatments were identical in appearance, taste, and packaging. In addition to participants, care providers, investigators, and outcomes assessors, the independent data monitoring committee and third-party statisticians involved in the primary data analysis were also masked to treatment assignments. The unblinding codes were securely held by a designated unmasked statistician who was not involved in the interim analyses or daily study conduct.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nimsai Herbal Group (Experimental): Participants in this arm received oral Nimsai Herbal (600 mg, one capsule per day) for 10 consecutive days.
  Interventions: Dietary Supplement: Nimsai Herbal
- Placebo Group (Placebo Comparator): Participants in this arm received oral placebo (identical in appearance, taste, and packaging to Nimsai Herbal) for 10 consecutive days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nimsai Herbal — Oral Nimsai Herbal is a novel botanical formulation, administered as one 600 mg capsule per day for a duration of 10 consecutive days. It is specifically designed to target the underlying venous congestion hypothesized by the War-Drill Model, aiming to promote hemorrhoid regression and symptom resolution.
  Arms: Nimsai Herbal Group
Dietary Supplement: Placebo — This intervention consisted of an oral placebo, formulated to be identical in appearance, taste, and packaging to Nimsai Herbal. It was administered as one capsule per day for 10 consecutive days to ensure blinding and serve as a control for comparison.
  Arms: Placebo Group

SUMMARY:
This study investigated a new understanding of hemorrhoid formation and evaluated a novel systemic treatment. For 200 years, hemorrhoids were conventionally understood as isolated swollen veins. However, our new "War-Drill Model" proposes that hemorrhoids are primarily caused by blood pooling (venous congestion) in the anal region, which then secondarily leads to vascular deformation. This congestion is hypothesized to arise from either underlying health issues ("War Mode") or natural physiological and hormonal changes ("Drill Mode"). We conducted a double-blind, placebo-controlled randomized controlled trial on 300 patients with Grade 2-3 hemorrhoids to evaluate the efficacy and safety of Nimsai Herbal. This study explores the potential for "War Mode" hemorrhoids to serve as an early warning sign for other serious underlying conditions and aims to validate a novel systemic therapeutic approach.

DETAILED DESCRIPTION:
The current understanding of hemorrhoid pathogenesis has remained largely unchanged for over two centuries, positing hemorrhoids primarily as isolated venous dilatations or prolapses. This traditional view, however, fails to adequately explain the high recurrence rates post-treatment, the limited efficacy of topical agents, and the often-debilitating symptomatology. Our extensive research, culminating in the "War-Drill Model" and the "Sine Qua Non Hypothesis," fundamentally challenges this conventional paradigm. We propose that hemorrhoids are not primarily structural abnormalities but rather a manifestation of underlying venous congestion, which then secondarily leads to vascular deformation and associated symptoms. This congestion acts as the indispensable (sine qua non) prerequisite for the development of both symptomatic and asymptomatic hemorrhoidal disease.

The "War-Drill Model" further categorizes this venous congestion based on its etiology:

War Mode Hemorrhoids: These are hypothesized to arise from chronic or passive venous congestion triggered by an underlying systemic or local inflammatory process or pathology. Examples include inflammatory bowel diseases (Crohn's disease, ulcerative colitis), anal fissures, rectal polyps, liver diseases causing portal hypertension, and various other systemic conditions affecting vascular flow or integrity. Crucially, "War Mode" hemorrhoids may serve as a critical "biological early-warning system," prompting investigations that could lead to the early diagnosis of up to 20 distinct and potentially severe internal diseases.

Drill Mode Hemorrhoids: These are hypothesized to be transient vascular engorgements resulting from physiological hormonal fluctuations, typically observed during periods of significant endocrine change such as adolescence, pregnancy, lactation, menopause, and andropause. These episodes are often self-limiting, resolving as hormonal balance stabilizes.

To validate a systemic therapeutic approach based on this new model, we conducted a double-blind, placebo-controlled, parallel-group Randomized Controlled Trial (RCT) (Protocol ID: NA-2024-01). The study enrolled 300 participants aged 18-70 years with endoscopically confirmed Grade 2-3 internal hemorrhoids and a history of symptoms for over 6 weeks. Participants were randomized to receive either Nimsai Herbal (a novel systemic botanical formulation, 600 mg daily) or an identical placebo for 10 consecutive days.

The primary outcome measure was hemorrhoid regression rate, defined as a reduction of at least one Goligher grade by Day 10, assessed via anoscopic examination and clinical evaluation. Secondary outcomes included incidence of adverse events. The study utilized the "Parola Phenomenon," a simple clinical maneuver designed by Atabiner, as part of patient assessment, aiming to differentiate War Mode from Drill Mode hemorrhoids.

ELIGIBILITY:
Inclusion Criteria:

Endoscopically confirmed Grade 2 or 3 internal hemorrhoids.

History of hemorrhoidal symptoms >6 weeks.

Age 18-70 years at the time of enrollment.

Provided written informed consent prior to any study-related procedures.

Willingness and ability to comply with all study procedures and follow-up visits.

Exclusion Criteria:

Grade 1 or 4 hemorrhoids.

Any known anorectal malignancy or suspicion of malignancy.

Pregnancy or lactation.

Known hypersensitivity or allergy to Nimsai Herbal components or placebo ingredients.

Significant systemic diseases (e.g., severe cardiovascular, renal, hepatic, or hematological disorders) that could affect study participation or safety.

Participation in another clinical trial within 30 days prior to screening.

Any condition that, in the opinion of the investigator, might compromise the safety of the participant or the integrity of the study data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cem Atabiner, Principal Investigator — Nimsai Academia
Locations (1):
- Nimsai Academia Clinical Research Center, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this article, after de-identification, will be available upon reasonable request to qualified researchers who submit a methodologically sound proposal. Data will be shared through a secure platform, subject to a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Individual participant data and supporting information will be available starting 6 months after the official publication of the primary manuscript in a peer-reviewed journal. The data will remain accessible indefinitely thereafter, or for as long as ethically and legally permissible under relevant data privacy regulations and institutional policies.
Access Criteria: Access to de-identified individual participant data (IPD) and supporting documentation (including the study protocol, statistical analysis plan, and informed consent form) will be granted to qualified researchers. Researchers must submit a methodologically sound and ethically approved research proposal that aligns with the original study's objectives or adds significant scientific value.
  Access will be provided through a secure, controlled-access platform, requiring a signed Data Use Agreement (DUA) between the requesting institution and Nimsai Academia. This agreement will outline strict terms for data use, confidentiality, and proper attribution, ensuring compliance with all applicable privacy regulations (e.g., GDPR, HIPAA equivalents). Data will be used solely for non-commercial scientific research purposes.
URL: https://kecioutdoor.com.tr/category/nimsai-academia/

REFERENCES:
- See also: Official website of Nimsai Academia, providing general information about the research institution and its activities. — https://kecioutdoor.com.tr/category/nimsai-academia/
- Available data/document: Study Protocol — https://kecioutdoor.com.tr/category/nimsai-academia/ — Access is subject to ethical approval of the research proposal by the Nimsai Academia Ethics Committee and the execution of a Data Use Agreement. Researchers must agree to use the data solely for scientific research and to respect participant privacy.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Group: Participants in this arm received oral placebo (identical in appearance, taste, and packaging to Nimsai Herbal) for 10 consecutive days.
  Nimsai Herbal: This intervention consisted of an oral placebo, formulated to be identical in appearance, taste, and packaging to Nimsai Herbal. It was administered as one capsule per day for 10 consecutive days to ensure blinding and serve as a control for comparison.
Period: Overall Study
Arm/Group | Nimsai Herbal Group | Placebo Group
Started | 150 | 150
Completed | 150 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants (N=300) were included in the baseline analysis population, as complete baseline data were obtained for all individuals.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimsai Herbal Group | Placebo Group | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 149 | 150 | 299
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.2 (12.3) | 45.7 (12.5) | 45.45 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 78 | 156
  Male | 72 | 72 | 144
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 150 | 150 | 300
Hemorrhoid Grade at Baseline [Count of Participants; unit: Participants] — Hemorrhoid severity was assessed at baseline using the Goligher classification: Grade 1 (no prolapse, may bleed); Grade 2 (prolapses with straining, spontaneous reduction); Grade 3 (prolapses with straining, manual reduction required); Grade 4 (permanently prolapsed, irreducible). Lower grades indicate less severe disease (e.g., Grade 1 < Grade 2 < Grade 3 < Grade 4). This study included participants with Grade 2 and Grade 3 hemorrhoids.
  Participants
    Grade 2 Hemorrhoids | 105 | 105 | 210
    Grade 3 Hemorrhoids | 45 | 45 | 90
Composite Severity Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — The Composite Severity Score is an aggregate measure assessing the overall severity of hemorrhoid symptoms. It is derived by summing individual scores from various primary symptoms, including pain, bleeding, itching, and prolapse, each rated on a Visual Analog Scale (VAS) from 0 to 10 (0 = no symptom, 10 = worst possible symptom). The total score ranges from 0 (no symptoms) to 40 (most severe symptoms across all assessed parameters). Higher scores indicate worse outcomes (greater symptom severity).
  units on a scale | 24.8 (6.7) | 24.5 (6.5) | 24.65 (6.6)
Overall Symptom VAS Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — The Overall Symptom VAS (Visual Analog Scale) Score is a patient-reported measure of global hemorrhoid symptom severity. Participants rated their overall symptom experience on a 10-point scale, where 0 represents "no symptoms" and 10 represents "worst possible symptoms." Higher scores indicate worse outcomes (greater overall symptom severity).
  units on a scale | 6.5 (1.9) | 6.4 (1.8) | 6.45 (1.85)
Participants with War Mode Hemorrhoids (via Parola Phenomenon) [Count of Participants; unit: Participants] — War Mode hemorrhoids were identified at baseline using the Parola Phenomenon, a clinical maneuver where participants are asked to contract their anal sphincter. An increase in throbbing sensation during contraction indicates War Mode, suggestive of underlying systemic or local pathology causing venous congestion. This measure reflects the proportion of participants presenting with War Mode hemorrhoids at study entry.
  Participants | 60 | 57 | 117
Diabetes (%) [Count of Participants; unit: Participants] | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Hemorrhoid Regression Rate
Description: Hemorrhoid regression was defined as a reduction of at least one Goligher grade or a ≥75% reduction in composite hemorrhoid severity score by Day 10. (The Goligher Classification of Hemorrhoids is a 4-point scale (Grade I to IV) used for hemorrhoid severity, where higher scores indicate worse disease.)
Time Frame: Day 10 (end of treatment period)
Population: All randomized participants who completed the study (Full Analysis Set).
Measure: Count of Participants; unit: Participants
Arm/Group | Nimsai Herbal Group | Placebo Group
Number analyzed (Participants) | 150 | 150
Participants | 117 | 33
Statistical Analysis 1: Comparison: Nimsai Herbal Group vs Placebo Group; Powered for 56% difference (80% power, alpha=0.05) to detect the anticipated difference in hemorrhoid regression rates between groups. The sample size of N=300 (150 participants per arm) was calculated based on an expected regression rate of 22% in the placebo group and 78% in the Nimsai Herbal group. This ensured sufficient statistical power for the primary efficacy analysis; Test type: Superiority; p < 0.001, Chi-squared — A priori statistical significance threshold for the primary endpoint was set at a two-sided alpha level of 0.05. No adjustment for multiple comparisons was applied to the primary outcome analysis, as it was the sole primary endpoint; Risk Difference (RD) = 56, 95% CI 2-sided [48 to 64] — The Risk Difference (RD) indicates the absolute difference in hemorrhoid regression rates between the Nimsai Herbal Group and the Placebo Group. Calculation: Nimsai Herbal (78%) - Placebo (22%) = 56%

ADVERSE EVENTS:
Time Frame: Adverse events were collected from randomization until the end of the study treatment period (Day 10), covering the entire intervention duration for each participant.
Description: Adverse events were systematically collected at each study visit and through participant spontaneous reports. Each event's severity and relationship to the study intervention were assessed by blinded investigators, ensuring robust and unbiased safety data collection.
Arm/Group | Nimsai Herbal Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/150
Other Adverse Events (participants affected / at risk) | 6/150 | 3/150
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimsai Herbal Group (N=150) | Placebo Group (N=150)
Mild GI discomfort (Gastrointestinal disorders) | 6 (6) | 3 (3) — Mild GI discomfort was the only reported non-serious AE, with incidence comparable between groups, likely unrelated to intervention.

LIMITATIONS AND CAVEATS:
This RCT focused on Grade 2-3 hemorrhoids; efficacy in Grade 1 and 4 needs further study. The short 14-day follow-up necessitates longer-term cohort studies for sustained effects. The Parola Phenomenon, though accurate, requires objective validation beyond clinical assessment. No formal blinding evaluation was conducted. Future research should explore potential genetic and microbiota interactions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (7):
  • Study Protocol: CASE REPORT FORMS (CRFs) (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT07034820/Prot_000.pdf
  • Study Protocol: INVESTIGATOR BROCHURE FOR NIMSAI HERBAL (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT07034820/Prot_001.pdf
  • Study Protocol: Study Flow Diagram (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT07034820/Prot_002.pdf
  • Study Protocol: In Vitro Mechanistic Evidence (Figures S2 and S3) (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT07034820/Prot_003.pdf
  • Study Protocol: Study Protocol ( Protocol NA-2024-01 ) (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT07034820/Prot_004.pdf
  • Statistical Analysis Plan (2021-10-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT07034820/SAP_005.pdf
  • Informed Consent Form (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT07034820/ICF_006.pdf